CLINICAL TRIAL: NCT03494569
Title: Phase I Study of Escalating Doses of Total Marrow and Lymphoid Irradiation (TMLI) Combined With Fludarabine and Melphalan as Conditioning for Allogeneic Hematopoietic Cell Transplantation in Patients With High-Risk Acute Leukemia or Myelodysplastic Syndrome
Brief Title: Total Marrow and Lymphoid Irradiation, Fludarabine, and Melphalan Before Donor Stem Cell Transplant in Treating Participants With High-Risk Acute Leukemia or Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17505; NCI-2018-00497 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17505 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia; Acute Myeloid Leukemia in Remission; Hematopoietic Cell Transplantation Recipient; Minimal Residual Disease; Myelodysplastic Syndrome; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Neoplasm, Residual; Myelodysplastic Syndromes | interventions — fludarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (TMLI, fludarabine, melphalan) (Experimental): Participants undergo TMLI BID on days -8 to -5, and receive fludarabine IV on days -4 to -2 and melphalan on day -2. Participants then undergo alloHCT on day 0.
  Interventions: Drug: Fludarabine; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Radiation: Total Marrow Irradiation

INTERVENTIONS:
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given as per City of Hope Standard Operating Procedure
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Radiation: Total Marrow Irradiation — Undergo TMLI

SUMMARY:
This phase I studies the side effects and best dose of total marrow and lymphoid irradiation when given together with fludarabine and melphalan before donor stem cell transplant in treating participants with high-risk acute leukemia or myelodysplastic syndrome. Giving chemotherapy, such as fludarabine and melphalan, and total marrow and lymphoid irradiation before a donor stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose/recommended phase II dose (MTD/RP2D) of total marrow and lymphoid irradiation (TMLI) with fixed doses of fludarabine and melphalan (FM100) as a preparative regimen in patients undergoing allogeneic hematopoietic stem cell transplantation (alloHCT) and who are not eligible for standard myeloablative regimens, with either a matched donor (Arm A) or a haploidentical donor (Arm B).

II. To describe toxicities attributable to TMLI by dose level in patients treated under this regimen.

SECONDARY OBJECTIVES:

I. To evaluate the safety of the regimen, at each dose level, by assessing the following: type, frequency, severity, attribution, time course and duration of adverse events, including acute/chronic graft versus host disease (GVHD), infection and delayed engraftment.

II. To investigate the temporal effect of bone marrow residual damage in alloHCT patients after TMLI/FM100.

III. To estimate overall survival (OS), event-free survival (EFS), cumulative incidence (CI) of relapse/progression, and non-relapse mortality (NRM) at 100 days, 1 year and 2 years.

IV. Assess minimal residual disease (MRD) from bone marrow aspirates on days 30, 100, and 180 post-transplant and describe its relation to TMLI dose level and patient disease status.

V. To evaluate effect of TMLI/FM100 conditioning on immune reconstitution after alloHCT in patients receiving stem cells from matched or haploidentical donors.

OUTLINE: This is a dose-escalation study of TMLI.

Participants undergo TMLI twice daily (BID) on days -8 to -5, and receive fludarabine intravenously (IV) on days -4 to -2 and melphalan on day -2. Participants then undergo alloHCT on day 0.

After completion of study treatment, participants are followed up twice weekly for 100 days, twice monthly for 6 months, and then monthly or yearly for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients with a histopathological confirmed diagnosis of hematologic malignancy in one of the following categories:

  * Acute myelogenous leukemia:

    * Patients with de novo or secondary disease in unfavorable risk group including poor risk cytogenetics according to National Comprehensive Cancer Network (NCCN) guidelines for AML i.e., monosomal karyotype, -5, 5q-, -7, 7q-, 11q23-non t (9;11), inv (3), t (3;3),t (6;9), t (9;22) and complex karyotypes (≥ 3 unrelated abnormalities), or all patient in intermediate risk groups accept patients with FLT3-NPM1+ disease
    * Patients with active disease
    * Patients with chemosensitive active disease
  * Acute lymphocytic leukemia:

    * Patients with de novo or secondary disease according to NCCN guidelines for ALL hypoploidy (< 44 chromosomes); t (v;11q23): MLL rearranged; t (9;22) (q34;q11.2); complex cytogenetics (5 or more chromosomal abnormalities); high white blood cell (WBC) at diagnosis (≥ 30,000 for B lineage or ≥ 50,000 for T lineage); iAMP21loss of 13q, and abnormal 17p
    * Patients with active disease
    * Patients with chemosensitive active disease
  * Myelodysplastic syndrome in high-intermediate (int-2) and high risk categories
* Patients ≥ 12 years and < 55 years are also included if they are not candidates for myeloablative conditioning regimens due to comorbidities
* Karnofsky or Lansky performance status of ≥ 70
* A pretreatment measured creatinine clearance (absolute value) of ≥ 60 ml/minute
* Patients must have a serum bilirubin ≤ 2.0 mg/dl
* Serum glutamic-oxaloacetic transaminase (SGOT) and serum glutamic-pyruvic transaminase (SGPT) ≤ 2.5 times the institutional upper limits of normal
* Ejection fraction measured by echocardiogram or multigated acquisition (MUGA) ≥ 50%
* Carbon monoxide diffusing capacity (DLCO) and forced expiratory volume FEV1 > 50% predicted
* PATIENT-SPECIFIC INCLUSION CRITERIA
* Patients should have discontinued all previous intensive therapy, chemotherapy or radiotherapy for 2 weeks prior to commencing therapy on this study

  * NOTE: low dose chemotherapy or maintenance chemotherapy given within 7 days of planned study enrollment is permitted; these include hydroxyurea, 6-meraptopurine, oral methotrexate, vincristine, oral etoposide, and tyrosine kinase inhibitors (TKIs); FLT-3 inhibitors can also be given up to 3 days before conditioning regimen
  * All patients with prior radiation treatment to the lung, liver, and kidney will be excluded; for other scenarios of prior radiation treatment, up to 2000 cGY at 2 gray Gy per day will be allowed; inclusion of patients with previous radiation exposure will be determined based on the radiation oncologist MD evaluation and judgment
* DONOR: Arm A: All candidates for this study must have an human leukocyte antigen (HLA) (A, B, C, and DR) identical sibling who is willing to donate primed blood stem cells (preferred) or bone marrow, or have a 10/10 (A, B, C, DR and DQ) allele matched unrelated donor; DQ or DP mismatch is allowed per discretion of the principal investigator
* DONOR: Arm B: The recipient must have a related donor genotypically HLA-A, B, C and DRB1 loci haploidentical to the recipient; no HLA matched sibling or matched unrelated donor is available; DSA is allowed with desensitization done if recommended by donor selection committee (DSC) per City of Hope (COH) standard operating procedures (SOP)
* DONOR: Both arms: All donors in both arms should be evaluated and approved by DSC

Exclusion Criteria:

* Having any uncontrolled illness including ongoing or active bacterial, viral or fungal infection
* Receiving any investigational agents or concurrent biological, intensive chemotherapy or radiation therapy for the previous 2 weeks from conditioning

  * NOTE: low dose chemotherapy or maintenance chemotherapy given within 7 days of planned study enrollment is permitted; these include: hydroxyurea, 6-meraptopurine, oral methotrexate, vincristine, oral etoposide, and tyrosine kinase inhibitors (TKIs), FLT-3 inhibitors can also be given up to 3 days before conditioning regimen
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to any in the regimen
* Patients with other malignancies are ineligible for this study, other than non-melanoma skin cancers
* The recipient has another medical problem or neurologic/psychiatric dysfunction which would impair his/her ability to be compliant with the medical regimen and to tolerate transplantation or would prolong hematologic recovery in which the opinion of the principal investigator would place the recipient at unacceptable risk
* Patients may not have had a prior autologous or allogeneic transplant
* Patients may not have received more than 3 prior lines of intensive chemotherapy, where the regimen intent was to induce remission
* In the opinion of the principal investigator (PI), the participant has a condition that will preclude them from complying with study treatment
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* All subjects must have the ability to understand and the willingness to sign a written informed consent; they are to give voluntary written informed consent before performance if any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care; cognitively impaired subjects will be included only if their guardian or legal representative agrees to sign the written informed consent
* DONOR: Donor selection for both arms must be approved by the donor selection committee
* DONOR: Evidence of active infection
* DONOR: Medical or physical reason which makes the donor unlikely to tolerate or cooperate with growth factor therapy or leukapheresis
* DONOR: Factors which place the donor at increased risk for complications from leukapheresis or granulocyte-colony stimulating factor (G-CSF) therapy could be harvested for bone marrow (BM) if safer for the donor and if approved by the principal investigator (PI)
* DONOR: Human immunodeficiency virus (HIV) positive

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-07-06 (Actual); Primary Completion 2026-09-08 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity | Up to 2 years
  Toxicity will be scored on both the Bearman scale and National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5 scale. Toxicity information recorded in each patient will include the type, severity, and the probable association with the study regimen. Tables will be constructed to summarize the observed incidence by severity and type of toxicity, and dose levels in each arm.

SECONDARY OUTCOMES:
Overall survival | From start of protocol therapy up to 2 years
  Participants are considered a failure for this endpoint if they die, regardless of cause. Survival estimates will be calculated using the Kaplan-Meier method.
Event-free survival | From start of protocol therapy up to 2 years
  Participants are considered a failure for this endpoint if they relapse/progress or die, regardless of cause. Survival estimates will be calculated using the Kaplan-Meier method.
Relapse/progression | From start of protocol therapy up to 2 years
  Death without relapse/progression is considered a competing risk.
Complete remission proportion | At day 30
Non-relapse mortality | Up to 2 years
  Participants are considered a failure for this endpoint if they die from causes other than disease relapse or progression.
Incidence of infection | Up to day 100 post-transplant
  Microbiologically documented infections will be reported by site of disease, date of onset, severity and resolution, if any. These data will be captured via case report form.
Incidence of toxicities/adverse events (AEs) | Up to 100 days post-transplant
  Toxicities that meet grade 3, 4, or 5 per the Bearman scale and CTCAE v 4.03 from day -9 to day -1, from day 0 to day +30, and again from day +31 to +100 post-transplant will be collected. Any AEs occurring from day -9 to day +30 will be followed until they resolve. Start and stop dates will also be recorded for any grade 4 neutropenia.
Neutrophil recovery | Up to 2 years
  This will be measured from stem cell infusion to the first to three consecutive days with neutrophil count greater than 0.5 x 10^9/l.
Acute graft versus host disease of grades 2-4 and 3-4 | Up to 100 days post-transplant
  Documented/biopsy proven acute graft versus host disease is graded according to National Institutes of Health (NIH) consensus staging. This measurement will be used to estimate the cumulative incidence.
Chronic graft versus host disease | Up to 2 years
  This will be scored according to NIH consensus staging and will be used to estimate the cumulative incidence.
CD4+, CD8+ and CD56+16+ | Up to 2 years
  Immunophenotyping of lymphocyte subsets will be determined by flow cytometry.
Bone marrow (BM) residual damage | Up to 2 years
  BM cellularity will be assessed using histology and clonogenic in vitro assays.
Immune reconstitution | Up to 2 years
  This will be monitored by flow cytometry analysis of peripheral blood mononuclear cells.

CONTACTS AND LOCATIONS:
Overall Officials: Monzr Al Malki, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States